CLINICAL TRIAL: NCT05991843
Title: Is it Possible to Measure an Adequate Respiration Rate Using Pressure Variation During HFNC
Brief Title: Respiratory Rate Measured by Pressure Variation During HFNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Mark Koning, Anesthesiologist-intensivist, principal investigator, Rijnstate Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL84438.091.23
Record Dates: First submitted 2023-07-30; First posted 2023-08-15 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Rate
Keywords: High Flow Nasal Cannula; Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study cohort (Experimental): The cohort of healthy volunteers, who will breath at three different respiratory rates, as guided by "normal", "slowly" and "rapid".
  Interventions: Behavioral: Instructions of breathing

INTERVENTIONS:
Behavioral: Instructions of breathing — Breathing normally, slowly and rapidly for 30 seconds with an open and a closed mouth.

SUMMARY:
Monitoring the respiratory rate is important during procedural sedation. Several methods of measuring the respiratory rate are available, but most are unreliable and the most reliable method (capnography) is not available during the use of High Flow Nasal Cannula (HFNC) oxygen. We hypothesize that measuring the pressure variation in the HFNC-circuit is a reliable method of measuring the respiratory rate.

An experimental study, using healthy volunteers that will breath in three guided respiratory rates, compares the measurements of respiratory rate by the pressure variation in the HFNC circuit with measurements of respiratory rate by an ECG-derived method and a manual count by an physician.

A secondary outcome will be the ability to measure the size of pressure difference, in order to determine its feasiblity to use it as a surrogate for tidal volume or respiratory effort.

DETAILED DESCRIPTION:
The healthy volunteers will be administered HFNC-oxygen and will be instructed to breath normally, rapidly and slowly for 30 seconds. This will be done at two HFNC flow rates (35 L/min and 70 L/min) and with an open and a closed mouth. During these 30 seconds the respiratory rate will be measured by pressure variation in the HFNC circuit, ECG-derived impedance difference and a manual count by a physician.

This will lead to 12 conditions, depending on HFNC flow (35 and 70 L/min), open or closed mouth and respiratory rate (normally, rapidly, slowly). The measurements of the respiratory rates wil be compared per HFNC flow and per open or closed mouth.

A secondary outcome will be the ability to measure the size of pressure difference, in order to determine its feasiblity to use it as a surrogate for tidal volume or respiratory effort.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* known neurodegenerative diseases
* Pregnancy
* Children (age <18)
* Upper airway obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Respiratory rate by pressure variation | 30 seconds
  Respiratory rate as measured by the pressure variation in the HFNC circuit.
Respiratory rate by manual count | 30 seconds
  Respiratory rate as measured by a physician
Respiratory rate by ECG-derived measurement | 30 seconds.
  Respiratory rate as measured by the ECG-derived impedance difference

SECONDARY OUTCOMES:
Pressure difference during breathing | 30 seconds.
  The pressure difference measured in the HFNC-circuit between inspiration and expiration in cmH2O as the mean value over the 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Mark V Koning, MD, PhD, Principal Investigator — Dept. of Anesthesiology and Critical Care, Rijnstate Hospital, Arnhem
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Available upon reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: Within 2 years
Access Criteria: Available upon reasonable request.

REFERENCES:
- [Result] Miechels J, Koning MV. Respiratory rate measurement by pressure variation in the high flow nasal cannula-system in healthy volunteers. J Clin Monit Comput. 2024 Dec;38(6):1397-1404. doi: 10.1007/s10877-024-01185-8. Epub 2024 Jun 12. PMID 38867018
- See also: Related Info — https://link.springer.com/article/10.1007/s10877-024-01185-8